CLINICAL TRIAL: NCT04497142
Title: Pilot Study of Perampanel on Peritumoral Hyperexcitability and Seizure Control in Newly Diagnosed High Grade Glioma
Brief Title: Effect of Perampanel on Peritumoral Hyperexcitability in HGG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Jong Woo Lee, MD PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-059; 2P50CA165962-06A1 (NIH)
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Glioma, Malignant; Surgery; Seizures
Keywords: Glioma; Surgery; Seizures
MeSH Terms: conditions — Glioma; Seizures | interventions — perampanel; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perampanel (Experimental): * Participants will take a predetermined first dose of perampanel on the day before their tumor surgery
  * During surgery, an approximately 4x6cm recording grid will be placed on the surface of the brain over the tumor, and brain activity around the tumor will be recorded for 10 minutes during surgery (Electrocorticography).
  * After surgery participants will take perampanel at a predetermined dose once a day for as long as they do not have serious side effects and their disease does not get worse, up to a maximum of 12 months. Participants will be provided a drug and seizure diary to document drug and seizure information and have monthly study visits either in clinic or by phone.
  Interventions: Drug: Perampanel
- Standard of Care (Active Comparator): * Participants will receive standard of care medication before surgery.
  * During surgery, an approximately 4x6cm recording grid will be placed on the surface of the brain over the tumor, and brain activity around the tumor will be recorded for 10 minutes during surgery (Electrocorticography).
  * After surgery participants will take standard of care medications as predetermined by their doctor. Participants will be provided a drug and seizure diary to document drug and seizure information and have monthly study visits either in clinic or by phone.
  * Participants will be followed up to 12 months after completing surgery.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Perampanel — Tablet taken orally 1x daily.
  Other Names: E2007; Fycompa
  Arms: Perampanel
Drug: Standard of Care — Predetermined standard of care drug and dosing
  Other Names: Standard treatment (typically the anti-seizure medication levetiracetam)
  Arms: Standard of Care

SUMMARY:
The purpose of this research study is to learn more about seizures in people with primary brain tumors. It will evaluate whether an antiseizure medication decreases hyperexcitability activity around tumors and prevents seizures.

The procedure and study drug involved in this study are:

* Electrocorticography
* Perampanel (Fycompa)

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining brain activity after taking perampanel.

The U.S. Food and Drug Administration (FDA) has approved perampanel as a treatment option for seizures. It has not been approved for the treatment of brain tumors. Recording of brain activity (electrocorticography) during surgery is an established clinical procedure, which will be performed for investigational purposes. This research study is studying brain recordings and perampanel treatment in participants with brain tumors for the following reasons:

* People with brain tumors commonly have seizures.
* Perampanel was developed as an anti-seizure medication, which works by blocking a signaling pathway between brain cells, mediated by AMPA receptors.
* Previous research has shown abnormal brain activity around tumors resulting from increased AMPA receptor activation.
* Perampanel is expected to decrease abnormal brain activity and prevent seizures by blocking AMPA receptor signaling.

This study involves two groups of participants, one group who receives the antiseizure medication perampanel, and the other group who receives the usual antiseizure medication (typically levetiracetam) at the time of surgery. Participants have the option to choose which group to participate if they have a preference.

The research study procedures include screening for eligibility, recording brain activity during surgery, and study treatment including evaluations and follow up visits. Participants will receive the study drug for as long as they do not have serious side effects and their disease does not get worse, up to a maximum of 12 months.

It is expected that about 20 people will take part in this research study.

The National Institute of Health (NIH) is supporting this study by providing funding for the research. Eisai Inc, a pharmaceutical company, is supporting this research study by providing the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have radiologic evidence of anaplastic astrocytoma or glioblastoma multiforme within 14 days of enrollment.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as ≥10 mm (≥1 cm) with CT or MRI. See Section 11 (Measurement of Effect) for the evaluation of measurable disease.
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Participants must have adequate organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
  * glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m2 (see Appendix B)
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* The effects of perampanel on the developing human fetus are unknown. For this reason and because some anti-seizure medications are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants with brain metastases due to confounding effects on the study objectives.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perampanel.
* Participants receiving any medications or substances that are moderate or strong inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Participants with uncontrolled intercurrent illness.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because perampanel is an anti-seizure agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with perampanel, breastfeeding should be discontinued if the mother is treated with perampanel.
* Participants with a history of suicide attempt or current active suicidal ideation with intent as defined by Columbia Suicide Severity Rating Scale (C-SSRS) type 4-5, due to the potential for suicidal ideation with the use of all anti-seizure medications.
* Participants who are unable to swallow pills.
* Participants with tumor associated seizures greater than one month before planned surgery.
* Participants currently receiving treatment with more than one anti-seizure medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Woo Lee, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Steven Tobochnik, MD at stobochnik@bwh.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Perampanel + Electrocorticography: Perampanel 6mg on day prior to resection, 4mg pre-op prior to resection, and 4mg daily until PD or up to 12 months. Intraoperative ECoG with 20 contact subdural grid performed for analysis of high frequency oscillation (80-500 Hz) rate.
- Standard of Care + Electrocorticography: Levetiracetam peri-operatively per standard of care. Intraoperative ECoG with 20 contact subdural grid performed for analysis of high frequency oscillation (80-500 Hz) rate.
Period: Overall Study
Arm/Group | Perampanel + Electrocorticography | Standard of Care + Electrocorticography
Started | 8 | 4
Completed | 7 | 4
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perampanel + Electrocorticography | Standard of Care + Electrocorticography | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 4 | 11
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Peritumoral HFO Rate
Description: Peritumoral hyperexcitability was measured by intraoperative electrocorticography (ECoG) high frequency oscillation (80-500 Hz) rate over 10 minutes within 1 cm of the contrast-enhancing margin at the time of initial glioma resection.
Time Frame: Peri-operative
Population: 1 participant (perampanel arm) was excluded from analysis after pathology revealed a non-glial tumor
Measure: Mean (Full Range); unit: HFOs per minute
Arm/Group | Perampanel + Electrocorticography | Standard of Care + Electrocorticography
Number analyzed (Participants) | 7 | 4
HFOs per minute | 2.5 [0 to 5.6] | 1.4 [0.4 to 3.0]

2. Secondary Outcome: Seizure-freedom
Description: Seizure-free rates were assessed from the time of initial glioma resection to radiographic tumor progression or up to a maximum of 12 months.
Time Frame: From time of initial surgery to PD or up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Perampanel + Electrocorticography | Standard of Care + Electrocorticography
Number analyzed (Participants) | 7 | 4
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: From the time of enrollment to PD or up to 12 months
Description: According to NCI CTCAE 5.0.
  Seizures were not considered adverse events per protocol as they were defined as a secondary outcome.
Arm/Group | Perampanel + Electrocorticography | Standard of Care + Electrocorticography
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 7/8 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel + Electrocorticography (N=8) | Standard of Care + Electrocorticography (N=4)
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0
Concentration impairment (Nervous system disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 3 | 2
Gait disturbance (General disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Hypersomnia (Nervous system disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination after planned interim analysis for futility. 1 participant (perampanel arm) was excluded from outcome analysis after pathology revealed a non-glial tumor, but was included in safety assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT04497142/Prot_SAP_001.pdf